CLINICAL TRIAL: NCT00683969
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter, 36-Week Trial to Assess the Efficacy and Safety of Adjunct Mycophenolate Mofetil (MMF) to Maintain or Improve Symptom Control With Reduced Corticosteroid in Subjects With Myasthenia Gravis
Brief Title: A Study to Assess the Effect of CellCept (Mycophenolate Mofetil) and Reduced Corticosteroids in Controlling Symptoms of Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Aspreva Pharmaceuticals (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WX17798; NCT00090636 (obsolete NCT alias)
Record Dates: First submitted 2008-05-19; First posted 2008-05-26 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-05

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: mycophenolate mofetil (CellCept)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mycophenolate mofetil (CellCept) — 1g bid for 36 weeks
  Arms: 1
Drug: placebo — po bid for 36 weeks
  Arms: 2

SUMMARY:
The efficacy and safety of CellCept (1g po, bid for 36 weeks) will be assessed in patients with myasthenia gravis receiving prednisone, or other corticosteroids. During the study, patients will undergo gradual corticosteroid dose reduction, if they respond to treatment. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18 to 80 years of age;
* diagnosis of myasthenia gravis;
* history of myasthenia weakness involving more than ocular (ie eye) or peri-ocular muscle;
* duration of myasthenia gravis symptoms (including ocular symptoms) <=10 years;
* prednisone dose >=20 mg/day (or equivalent alternate-day dose) for >=4 weeks.

Exclusion Criteria:

* female patients who are pregnant, breastfeeding, or lactating;
* regularly scheduled plasma exchange (PE) or intravenous immunoglobulin (IVIG) treatment, or PE or IVIG treatment within 2 weeks prior to randomization;
* any prior clinically significant use of CellCept or other immunosuppressive therapy (except corticosteroids), or within 8 weeks prior to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2004-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects reaching responder status | Week 36

SECONDARY OUTCOMES:
Time to start of response | Event driven
Mean and median prednisone dose and cholinesterase inhibitor dose | Week 36
Adverse events, lab parameters, vital signs | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche, 973-235-5000
Locations (41):
- United States (10):
  - Sun City, Arizona
  - Sacramento, California
  - Miami, Florida
  - Kansas City, Kansas
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Upland, Pennsylvania
  - Dallas, Texas
  - Galveston, Texas
- Canada (2):
  - Edmonton, Alberta
  - London, Ontario
- France (2):
  - Bordeaux
  - Nice
- Germany (4):
  - Düsseldorf
  - München
  - Regensburg
  - Tübingen
- India (3):
  - Hyderabad
  - Mumbai
  - New Delhi
- Jerusalem, Israel
- Italy (3):
  - Milan
  - Roma
  - San Donato Milanese
- Mexico City, Mexico
- Netherlands (3):
  - Leiden
  - Maastricht
  - Rotterdam
- Russia (3):
  - Kazan'
  - Moscow
  - Nizhniy Novgorad
- Belgrade, Serbia and Montenegro
- Spain (2):
  - Barcelona
  - Madrid
- Ukraine (3):
  - Kharkiv
  - Kiev
  - Zaporizhzhya
- United Kingdom (3):
  - Liverpool
  - Oxford
  - Salford

REFERENCES:
- [Derived] Sengupta M, Cheema A, Kaminski HJ, Kusner LL; Muscle Study Group. Serum metabolomic response of myasthenia gravis patients to chronic prednisone treatment. PLoS One. 2014 Jul 17;9(7):e102635. doi: 10.1371/journal.pone.0102635. eCollection 2014. PMID 25032816